CLINICAL TRIAL: NCT05014906
Title: Efficacy of 45mg Oral Minocycline (Solodyn) and 45mg Oral Minocycline (Solodyn) Plus 15% Azelaic Acid (Finacea) in the Treatment of Acne Rosacea
Brief Title: Efficacy of Oral Minocycline (Solodyn) and Oral Minocycline (Solodyn) Plus Azelaic Acid (Finacea) for Acne Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatology Specialists Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ROS001
Record Dates: First submitted 2013-11-22; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Rosacea
Keywords: rosacea
MeSH Terms: conditions — Rosacea | interventions — Minocycline; azelaic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- minocycline, azelaic acid (Active Comparator): minocycline vs minocycline in comination with 15% azelaic acid for treatment of rosacea
  Interventions: Drug: Minocycline 45 MG; Drug: Azelaic acid
- azelaic acid (Experimental): 45 mg oral minocycline vs 45 mg oral minocycline plus 15% azelaic acid in the treatment of facial rosacea
  Interventions: Drug: Minocycline 45 MG; Drug: Azelaic acid

INTERVENTIONS:
Drug: Minocycline 45 MG — 45 mg oral minocyclineonce daily vs 45mg oral minocycline once daily in combination with use of 15% azelaic acid
  Other Names: Solodyn
Drug: Azelaic acid — 45 mg oral minocyclineonce daily vs 45mg oral minocycline once daily in combination with use of 15% azelaic acid
  Other Names: finacea

SUMMARY:
Rosacea is one of the most commonly occurring dermatoses treated by dermatologist today. Rosacea is an inflammatory condition of the skin presenting as flushing and or blushing along with redness, swelling, telangiectasia, and acne lesions. Minocycline has shown beneficial in the treatment of inflammatory acne lesions in patients with rosacea. This study is to evaluate the efficacy and tolerability of minocycline (Solodyn) alone versus minocycline (Solodyn) in combination with azelaic acid 15%(Finacea) in the treatment of rosacea.

DETAILED DESCRIPTION:
This is a multicenter, randomized, outpatient, Investigator-blind study of minocycline 45 mg and minocycline 45 mg plus 15% azelaic acid for the treatment of rosacea.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older with clinical diagnosis of rosacea
* must have 10-40 facial inflammatory lesions and less than 2 nodules
* women of child bearing potential must be non lactating
* must have negative urine pregnancy test
* must use effective form of birth control

Exclusion Criteria:

* The use of systemic antibiotics within 30 days of study start
* the use of topical medications within 14 - 30 days of study start depending on type of topical medication
* Patients with known sensitivity to tetracyclines
* Patients who have had gastric bypass surgery or are considered achlorhydric
* Patients taking drugs known as photosensitizers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Efficacy analysis of the 12-week reduction in total lesion count | 12 weeks
  The goal of analysis is to assess evidence of overall effect of 45mg minocycline and overall effect of 45 mg minocycline plus 15% azelaic acid in therapy of patients with acne rosacea.

SECONDARY OUTCOMES:
Efficacy analysis of the12 week reduction in IGA (Investigators Global Assessment) per treatment group | 12 Weeks
  Summary of the 12-week reduction in IGA for the full sample, by treatment group
Efficacy analysis of the 12-week reduction in CEA (Clinical Erythema Assessment) per treatment group | 12 Weeks
  Summary of the 12 week reduction in CEA for the full sample, by treatment group

OTHER OUTCOMES:
Tolerability of treatment per group | 12 Week
  Summary of adverse events suspected as related to study medication per treatment group

CONTACTS AND LOCATIONS:
Overall Officials: James M Jackson, MD, Principal Investigator — Dermatology Specialists
Locations (1):
- Dermatology Specialists, Louisville, Kentucky, United States